CLINICAL TRIAL: NCT03444220
Title: Reduce Disease Activity in Systemic Sclerosis by Transplantation of an Anaerobically Cultivated Human Intestinal Microbiota, a Controlled Interventional Pilot Trial
Brief Title: Gut Microbiota Transplantation in Systemic Sclerosis
Acronym: ReSScue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anna-Maria Hoffmann-Vold, Principle Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/1529
Record Dates: First submitted 2018-02-13; First posted 2018-02-23 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACHIM (Active Comparator): Anaerobically Cultivated Human Intestinal Microbiota
  Interventions: Biological: Anaerobically Cultivated Human Intestinal Microbiota
- Placebo (Placebo Comparator): Anaerobically Cultivated medium
  Interventions: Biological: Anaerobically Cultivated medium

INTERVENTIONS:
Biological: Anaerobically Cultivated Human Intestinal Microbiota — 30ml ACHIM will be administrated at week 0 and 2 with 14 days apart
  Arms: ACHIM
Biological: Anaerobically Cultivated medium — 30ml medium will be administrated at week 0 and 2 with 14 days apart
  Arms: Placebo

SUMMARY:
Systemic Sclerosis (SSc) is a progressive multi-organ disorder with high disease burden. Life expectancy in SSc is reduced by 25-40 years, mainly due to cardiopulmonary and gastro-intestinal (GI) disease involvement; and a very poor response to available treatment. Aiming to improve treatment for SSc, the ReSScue project will determine the therapeutic potential of standardized, cultivated gut microbiome transplantation (GMT), and assess the mechanisms by which this novel intervention strategy works. This approach is rationalized by studies indicating that skewed gut microbiomes could act as major, environmental risk factors in SSc; and thereby be rational targets for therapeutic manipulation. ReSScue is set up as a 4 months randomized double blind trial involving the University Hospital in Oslo. Trial participants will be recruited from the population-based, nationwide SSc cohort. Intervention will be by GMT or placebo. Primary end point is changes in SSc-related GI parameters , while secondary outcomes include safety, explorative clinical parameters, changes in oral, skin and gut microbiomes, and in immune cell phenotypes.

DETAILED DESCRIPTION:
This is a randomized, double blind clinical trial testing intervention by standardized GMT. The study cohort will include 10 SSc patients with GI symptoms. Evaluation of end points is at 16 weeks. The trial is set up with six study visits. Patient recruitment, eligibility screening and retrieval of informed consent will be performed at OUS before inclusion. At visit 1, and 6 patients will undergo clinical examination, PFTs, at all visits clinical examination and sampling of biological material.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the 2013 SSc classification criteria
* Objective GI involvement and provide informed consent.

Exclusion Criteria:

* Severe organ dysfunction (and risk of procedure related complications
* Recent exposure to antibiotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Clinical SSc-related GI parameters | The change in the UCLA GIT score from baseline to week 16 will be evaluated.
  The investigators apply a patient-reported outcome measure; the validated UCLA Scleroderma Clinical Trial Consortium GIT 2.0 (UCLA GIT score 2.0) Instrument.
  The instrument includes seven multi-item scales: diarrhea, reflux, distention/bloating, fecal soilage, constipation, emotional well-being, and social functioning. Items are scored on a 0-3 range, and a lower value indicates a better health related quality of life. The Total GIT Score is a composite score that includes the total sum of all subgroups except constipation divided by 6. The Total GIT Score ranges from 0-3, and a lower value indicates a better health related quality of life.

SECONDARY OUTCOMES:
Clinical SSc activity | The investigators will assess all the SSc disease activity index measures at study start and week 16 .
  Explore the effect of GMT on known clinical outcome measures. The investigators base these assessments on the validated SSc disease activity index which includes a set value for active disease and a definition of change.
Gut microbiome composition changes | The investigators will assess the gut microbiome weekly from study start to week 16.
  It is unknown how the gut microbiome composition changes after GMT and how long these changes persist. We will investigate these aspects, as well as the mechanisms by which ACHIM exert its effects. Specifically, the investigators will address how the intestinal IgA binding to gut commensals and other bacteria is regulated.
Incidence of Treatment-Emergent Adverse Events (Safety) | Explore safety of GMT intervention at each study visit (week 0, 2, 4, 8,12 and 16)
  We define an adverse event as any untoward medical occurrence that may arise during the study period. The study investigator will fill out a safety form at each study visit (week, 0, 2, 4, 8, 12 and 16). The following questions will be asked: Hospital admission or contact with primary physician since last visit and reason why. Diarrhea, constipation, stomach pain, nausea, vomiting or fever since last study visit. Use of antibiotics since last visit.
Tissue architecture changes | The investigators will analyse tissue architeure in the gut at week 0. 2 and 16. The skin tissue archtecture at week 0 and 16. The immune cell distribution in blood at week 0, 2, 4, 8, 12 and 16.
  Explore effects of GMT on tissue architecture in gut and skin, and on immune cell distribution in blood.
Clinical SSc-related GI parameters | The change in the UCLA GIT score from baseline will be evaluated at each study visit (week 0,2,4,8 and 12).
  The investigators apply a patient-reported outcome measure; the validated UCLA Scleroderma Clinical Trial Consortium GIT 2.0 (UCLA GIT score 2.0) Instrument.
  The instrument includes seven multi-item scales: diarrhea, reflux, distention/bloating, fecal soilage, constipation, emotional well-being, and social functioning. Items are scored on a 0-3 range, and a lower value indicates a better health related quality of life. The Total GIT Score is a composite score that includes the total sum of all subgroups except constipation divided by 6. The Total GIT Score ranges from 0-3, and a lower value indicates a better health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Maria Hoffmann-Vold, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Strahm N, Didriksen H, Fretheim H, Molberg O, Midtvedt O, Farstad IN, Midtvedt T, Lundin KEA, Aabakken L, Blyszczuk P, Distler O, Kania G, Hoffmann-Vold AM. Effects of faecal microbiota transplantation on the small intestinal mucosa in systemic sclerosis. Rheumatology (Oxford). 2023 Aug 1;62(8):2918-2929. doi: 10.1093/rheumatology/kead014. PMID 36688692